CLINICAL TRIAL: NCT06013176
Title: Behavioral Economic Strategies to Improve PRO Adherence
Acronym: BEST-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 34923; P50CA244690 (NIH); 852748 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will be identified pragmatically and will be independently randomized to study arms using a three-arm design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual practice (No Intervention): This arm will consist of encounter-based PRO monitoring, in which patients have an opportunity to complete PRO questionnaires via patient portal in advance of clinical encounters or via tablet during clinical encounters. While clinicians will be encouraged to view and discuss PROs with patients during clinical encounters, they will not be prompted to do so in real-time, nor will there be alerts for escalating symptoms.
- Encounter-based PRO monitoring (Experimental): Encounter-based PRO monitoring (usual practice) plus patient reminders and triage nurse alerts
  Interventions: Other: Encounter-based PRO monitoring
- Remote PRO monitoring (Experimental): Remote PRO monitoring plus patient reminders and triage nurse alerts
  Interventions: Other: Remote PRO monitoring

INTERVENTIONS:
Other: Encounter-based PRO monitoring — This arm consists of usual practice plus the addition of patient reminders to complete PRO questionnaires and triage nurse alerts for severe symptoms. Patient reminders will be operationalized through the Epic patient portal. Triage nurse alerts will be routed to Epic symptom management pools in response to a patient reporting moderate or severe symptoms. Patients will have the opportunity to decline or opt-out of triage nurse support. Clinical interventions stemming from triage nurse alerts will be up to the discretion of clinical teams - i.e., clinical responses will be neither prescriptive nor mandatory. Notably, the entry point for triage nurse alerts (i.e., Epic symptom management pools), as well as resultant clinical responses, are existing standard operating procedures/practices for patients reporting symptoms by phone.
  Arms: Encounter-based PRO monitoring
Other: Remote PRO monitoring — This arm will consist of weekly PRO questionnaires administered via the patient portal, de-linked from clinical encounters. Patient reminders will be operationalized through the Epic patient portal. Triage nurse alerts will be routed to Epic symptom management pools in response to a patient reporting moderate or severe symptoms. Patients will have the opportunity to decline or opt-out of triage nurse support. Clinical interventions stemming from triage nurse alerts will be up to the discretion of clinical teams - i.e., clinical responses will be neither prescriptive nor mandatory. Notably, the entry point for triage nurse alerts (i.e., Epic symptom management pools), as well as resultant clinical responses, are existing standard operating procedures/practices for patients reporting symptoms by phone.
  Arms: Remote PRO monitoring

SUMMARY:
The main purpose of this research study is to evaluate the implementation and effectiveness of patient- and nurse-directed strategies across in-clinic and remote patient reported outcome (PRO) monitoring settings, using a three-arm pragmatic cluster randomized controlled trial. Additionally, the goal is to evaluate moderators of implementation effects on PRO monitoring.

Eligible patients will be randomized independently to: (1) usual practice (i.e., encounter-based PRO administration via patient portal or tablet); (2) encounter-based PRO monitoring with patient reminders and nurse alerts; or (3) remote PRO monitoring with patient reminders and nurse alerts. The investigators hypothesize that nudges to patients and alerts to nurses will improve patient-level PRO completion and clinician-level PRO engagement.

DETAILED DESCRIPTION:
Routine PRO monitoring is an evidence-based practice that improves patient outcomes. Patients with cancer commonly experience symptoms which go unrecognized by clinical teams up to half of the time. PROs are a powerful tool to bridge this gap, amplifying the patient experience and improving communication between patients and clinicians. A seminal clinical trial was conducted in which weekly PRO symptom assessments with care team alerts led to reduced care utilization, improved quality of life, and lengthened overall survival among patients receiving active treatment for advanced solid tumors. Subsequent randomized trials have corroborated the quality of life and survival advantages of PRO monitoring in other cancer populations and practice settings.

Real-world adherence to PRO monitoring is lower than in seminal clinical trials, with potential racial/ethnic disparities. Multilevel barriers to PRO implementation exist at the patient, clinician, practice, and system levels. While patient adherence to PRO monitoring in seminal trials ranged from 70 to 90 percent, real-world adherence is much lower and more variable. Our preliminary research demonstrates that in a large, multi-site rollout of PRO monitoring, mean patient-level adherence was less than 50 percent. Moreover, compared to non-Hispanic White patients, Black and Hispanic patients were 9% and 4% less likely to complete PRO questionnaires, respectively, but more likely to report more severe symptoms. These results highlight that historically marginalized subgroups may benefit less from current methods of PRO administration, potentially reinforcing existing disparities in symptom management if not remediated.

This will be the first study to apply behavioral economic strategies to align clinicians and patients in achieving sustained patient-level PRO adherence, and addresses limitations of current PRO approaches. Current approaches to PRO collection are limited by: (1) suboptimal clinician engagement, (2) encounter-based assessments which preclude longitudinal monitoring of PROs outside of the clinic, and (3) insufficient automated effectors actively linking reported symptoms with clinical response. This proposal addresses these limitations by employing behavioral strategies directly targeting clinician engagement, utilizing novel electronic remote monitoring methods to maximize real-time PRO capture, and linking these with pathway-driven automated effectors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must initiate a new line of systemic cancer therapy (i.e., intravenous chemotherapy or immunotherapy) at a participating Implementation Lab site

Exclusion Criteria:

- Patient opts out of pragmatic research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Parikh, MD, Principal Investigator — University of Pennsylvania; Emory University; Samuel Takvorian, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Practice | Encounter-based PRO Monitoring | Remote PRO Monitoring
Started | 171 | 144 | 161
Completed at least one questionnaire | 115 | 106 | 118
Completed | 171 | 144 | 161
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Practice | Encounter-based PRO Monitoring | Remote PRO Monitoring | Total
Number analyzed (Participants) | 171 | 144 | 161 | 476
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 51 | 64 | 184
  >=65 years | 102 | 93 | 97 | 292
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 58 | 55 | 179
  Male | 105 | 86 | 106 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 161 | 135 | 154 | 450
  Not Hispanic or Latino | 4 | 6 | 2 | 12
  Unknown or Not Reported | 6 | 3 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 5 | 7 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 44 | 27 | 36 | 107
  White | 110 | 102 | 104 | 316
  More than one race | 1 | 3 | 0 | 4
  Unknown or Not Reported | 9 | 5 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 171 | 144 | 161 | 476

OUTCOME MEASURES:

1. Primary Outcome: PRO Adherence
Description: The primary outcome will be PRO adherence, measured at the patient level as the proportion of expected PRO questionnaires completed per patient.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: pct. assigned questionnaires completed
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
pct. assigned questionnaires completed | 50.0 [43.9 to 56.1] | 56.9 [50.4 to 63.4] | 34.9 [29.8 to 40.0]

2. Secondary Outcome: Percent of Patients With at Least One Note Documenting PROs During Study Period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
Participants | 67 | 82 | 96

3. Secondary Outcome: Percent of Patients With at Least One Note Documenting PROs Per Month During Study Period
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
Participants | 20 | 16 | 32

4. Secondary Outcome: Time to Alert Response (for Arms 2 and 3 Only)
Time Frame: 3 months
Population: Clinical teams documented responses to patients' questionnaire submissions within the electronic health record.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: Responses to questionnaire submissions
Arm/Group | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 144 | 161
Number analyzed (Responses to questionnaire submissions) | 113 | 176
days | 1.24 (1.06) | 1.20 (1.01)

5. Secondary Outcome: Percent of Patients Who Trigger an Alert for Triage Nurses (for Arms 2 and 3 Only)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 144 | 161
Participants | 71 | 84

6. Secondary Outcome: Acute Care Utilization
Description: Percent of patients with an emergency department visit or hospitalization
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
Participants | 48 | 45 | 51

7. Secondary Outcome: Treatment Modifications
Description: Percent of patients with a treatment modification
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
Participants | 43 | 35 | 29

8. Secondary Outcome: Duration of Therapy
Description: Average duration of therapy during the study period
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual practice | Encounter-based PRO monitoring | Remote PRO monitoring
Number analyzed (Participants) | 171 | 144 | 161
days | 56.82 (31.67) | 55.94 (33.91) | 53.66 (32.62)

ADVERSE EVENTS:
Time Frame: 12 weeks following enrollment
Arm/Group | Usual Practice | Encounter-based PRO Monitoring | Remote PRO Monitoring
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/144 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/144 | 0/161
Other Adverse Events (participants affected / at risk) | 0/171 | 0/144 | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT06013176/Prot_SAP_000.pdf